CLINICAL TRIAL: NCT06456437
Title: Ischemic Post-conditioning in the Treatment of Acute Ischemic Stroke--a Multicenter, Prospective Cohort Study
Brief Title: Ischemic Post-conditioning in the Treatment of Acute Ischemic Stroke
Status: Recruiting | Type: Observational
Sponsor: Ming Wei (Other)
Responsible Party: Sponsor-Investigator, Ming Wei, Director, Head of Neurosurgery, Principal Investigator, Clinical Professor, Tianjin Huanhu Hospital
Organization: Tianjin Huanhu Hospital (Other)
Other Study IDs: TJHH-2023-WM26
Record Dates: First submitted 2024-05-30; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Acute Ischemic Stroke; Large Vessel Occlusion; Intracranial Artery Occlusion With Cerebral Infarction; Endovascular Treatments
Keywords: Endovascular treatments; Acute ischemic stroke; Retrieved clots; Ischemic Post-conditioning; Stroke etiology
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — Thrombosis specimens；Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Post-ischemic adaptation to combined endovascular therapy
  Interventions: Device: Post-conditioning Balloon dilation and contraction
- Endovascular therapy alone

INTERVENTIONS:
Device: Post-conditioning Balloon dilation and contraction — The balloon was filled at a pressure of no more than 4 atm at the original occlusion of the vessel to block blood flow for 2 minutes (confirmed by angiography), and then contracted to reperfuse the blood flow for 2 minutes, and the above steps were repeated 4 times to complete the in situ ischaemic post-acclimatisation intervention.
  Groups: Post-ischemic adaptation to combined endovascular therapy

SUMMARY:
Post-ischemic adaptation is a physical brain protective treatment strategy in which an ischemic event in an organ or tissue is treated and blood flow is restored, and an ischemic stimulus is given to local tissues to induce the production of anti-ischemic damage factors and reduce the damage associated with reperfusion therapy . Relevant basic studies have confirmed that post-ischemic adaptation can reduce infarct volume and promote neurological function recovery in animal models of cerebral infarction. Therefore, it may be beneficial to the recovery of neurological function in patients with acute ischemic stroke undergoing mechanical thrombus extraction.

Based on the above background, the use of a balloon to repeatedly dilate-contract at the original occlusion site after revascularization to block and restore arterial flow may be an effective cerebroprotective treatment for patients with large-vessel occlusion who undergo thrombolysis. However, can this approach be safely used in patients with acute ischemic stroke treated with thrombolysis? What is the protocol for the length of time patients can tolerate post-ischemic adaptation? The application of this method in the treatment of acute ischemic stroke will be explored in this study.

DETAILED DESCRIPTION:
Stroke has become the second leading cause of death in the world and the first cause of death and disability in adults in China; among them, ischemic stroke (AIS) accounts for about 80% of all strokes, and is the most important type of stroke . Ischemic stroke is usually caused by acute occlusion of cerebral blood vessels, therefore, opening the occluded blood vessels is the key to its treatment; at present, intravenous thrombolysis and endovascular mechanical thrombolysis are recommended by domestic and international guidelines for recanalization of blood vessels, and they have become the most effective treatment measures for ischemic stroke . However, due to the short therapeutic time window (<4.5 hours) and low recanalization rate of large vessel occlusion (less than 20%) of intravenous thrombolysis, endovascular mechanical thrombolysis is increasingly favored because of its long therapeutic time window, high recanalization rate of large vessel occlusion, and other advantages . However, although mechanical thrombolysis has a high rate of revascularization, the clinical prognosis of patients is not satisfactory, and both domestic and international studies have found that among patients treated with mechanical thrombolysis, the percentage of disability-free at 3 months is less than 30%, while the rate of death and disability is as high as more than 70% . The ischemia-reperfusion injury that occurs after revascularization may be the root cause of patients' still unsatisfactory prognosis . Therefore, trying to reduce ischemia-reperfusion injury after opening the occluded vessel to further improve the prognosis of patients is a scientific problem that needs to be solved urgently nowadays.

At present, scholars at home and abroad agree that effective neuroprotective therapy based on revascularization is expected to be an important treatment method to further improve the prognosis of patients with AIS, but there is no conclusion on how revascularization should be combined with neuroprotective therapy ; moreover, although a large number of studies have been carried out on neuroprotective therapy for acute ischemic stroke and hundreds of measures have been confirmed to have neuroprotective effects by animal experiments, the neuroprotective effects of such measures are not yet known. In addition, although a large number of studies have been conducted on neuroprotective therapy for acute ischemic stroke, and hundreds of measures have been demonstrated to be neuroprotective by animal experiments, there are still no clinically available neuroprotective measures .

Post-ischemic adaptation is a physical brain protective treatment strategy in which an ischemic event in an organ or tissue is treated and blood flow is restored, and an ischemic stimulus is given to local tissues to induce the production of anti-ischemic damage factors and reduce the damage associated with reperfusion therapy . This method has been widely studied in the field of coronary heart disease rescue, and the results suggest that in situ ischemic post-adaptation immediately after coronary revascularization can safely and effectively reduce ischemia-reperfusion myocardial injury, reduce the size of myocardial infarction, and improve clinical prognosis . The process of mechanical thrombolysis for acute ischemic stroke is similar to that of emergency recanalization for acute coronary syndromes, and relevant basic studies have confirmed that post-ischemic adaptation can reduce infarct volume and promote neurological function recovery in animal models of cerebral infarction. Therefore, it may be beneficial to the recovery of neurological function in patients with acute ischemic stroke undergoing mechanical thrombus extraction.

Based on the above background, the use of a balloon to repeatedly dilate-contract at the original occlusion site after revascularization to block and restore arterial flow may be an effective cerebroprotective treatment for patients with large-vessel occlusion who undergo thrombolysis. However, can this approach be safely used in patients with acute ischemic stroke treated with thrombolysis? What is the protocol for the length of time patients can tolerate post-ischemic adaptation? The application of this method in the treatment of acute ischemic stroke will be explored in this study.

ELIGIBILITY:
Inclusion Criteria:

* 1)Ischemic stroke confirmed by CT or MRI of the head;
* 2) Large vessel occlusion confirmed by CTA or MRA of the head, including: intracranial internal carotid artery (ICA), middle cerebral artery (MCA M1/M2), anterior cerebral artery (ACA A1/A2), basilar artery (BA), vertebral artery (VA), and posterior cerebral artery (PCA P1/P2);
* 3) Recanalization of the occluded vessel at eTICI grade 2b/3 as confirmed by DSA after thrombectomy;
* 4)The patient/legally authorized representative has signed an informed consent form.

Exclusion Criteria:

* 1) Inability to perform an MRI or CT scan for any reason;
* 2）The patient has any condition that would interfere with neurologic assessment or psychiatric disorders;
* 3）Stroke onset with seizures resulted in the inability to obtain an accurate NIHSS baseline;
* 4）Pregnancy
* 5）Other serious, advanced or terminal illness;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute cerebral infarction receiving endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Infarct volume at 24(-6/+12) h postoperatively | 24 (-6/+12) h postoperatively
  Infarct volume at 24(-6/+12) h postoperatively (CT/DWI, preferred DWI)

SECONDARY OUTCOMES:
Change in final cerebral infarct volume relative to baseline at 24 (-2/+12) hours postoperatively on CT/MR | 24 hours after thrombectomy
  Change in final cerebral infarct volume relative to baseline at 24 (-2/+12) hours postoperatively on CT/MR
Postoperative 90 d mRS score (0-2 vs 3-6) | 90 days after thrombectomy
  Percentage of mRS scores 0-2 vs 3-6 at 90 d postoperatively
Postoperative 90 d mRS score (0-3 vs 4-6) | 90 days after thrombectomy
  Percentage of mRS scores 0-3 vs 4-6 at 90 d postoperatively
Distribution of mRS scores at 90 d postoperatively | 90 days after thrombectomy
  Distribution of mRS（modified Rankin scale）scores at 90 d postoperatively
NIHSS score at 24 h postoperatively | 24 hours after thrombectomy
  NIHSS(National Institute of Health stroke scale) score at 24 h postoperatively
Proportion of patients with a good prognosis early after treatment | 24 hours after thrombectomy
  Decrease in NIHSS score ≥ 8 or NIHSS score of 0-2 in 24 (-2/+12) hours
NIHSS score at 7 d postoperatively/discharge | 7 days after thrombectomy/time of discharge
  NIHSS(National Institute of Health stroke scale) score at 7 d postoperatively/discharge
Vascular recanalization | 24 hours after thrombectomy
  Postoperative revascularisation assessed by CTA/MRA/DSA using Arterial Occlusive Lesion (AOL) grading at 24 (-2/+12) hours postoperatively； Postoperative revascularisation assessed by CTA/MRA/DSA using modified Thrombolysis In Cerebral Infarction(mTICI) grading at 24 (-2/+12) hours postoperatively； Application of bedside TCD for assessment of revascularisation
Haemodynamic assessment within 24 h postoperatively (confirmed by CTA, MRA, DSA or TCD) | 24 hours after thrombectomy
  This was defined as an exploratory outcome: primary measures included CT or MR perfusion, dynamic contrast contrast-enhanced magnetic resonance (DCE MRI) or permeability surface (PS) detection of the blood-brain barrier.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Wei, doctorate, Principal Investigator — Tianjin Huanhu Hospital
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China